CLINICAL TRIAL: NCT00694395
Title: Decision Making Process in Patients With Symptoms of Acute Ischemic Stroke Why do They Delay in Seeking Medical Help? A Qualitative Study
Brief Title: A Qualitative Study of Delays in Hospital Admission in Patient With Acute Stroke
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Fu Jen Catholic University (Other)
Responsible Party: Dr. Lung, Chan, Far Eastern Memorial Hospital
Other Study IDs: 95013
Record Dates: First submitted 2008-06-05; First posted 2008-06-10 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2006-07

CONDITIONS: Acute Ischemic Stroke
Keywords: Qualitative study; stroke; 20 patients, Family or caregivers; acute ischemic stroke; delayed to receive thrombolytic therapy.
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To identify the circumstance during decision making processes to seek medical help in patients with symptoms of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed acute ischemic stroke by brain image and were able to communicate in Mandarin or Taiwanese.

Exclusion Criteria:

* patients who had cerebral hemorrhage, aphasia, cognitive dysfunction or severe stroke with unstable vital sign.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients admitted to hospital due to acute ischemic stroke and were delayed to receive thrombolytic therapy. Family or caregivers who had involved in the process of decision making were also invited to the interview.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2006-08; Primary Completion 2007-05 (Actual); Study Completion 2007-07 (Actual)